CLINICAL TRIAL: NCT06971419
Title: FOllow-Up of LOW-Acuity Patients After REdirection From the Emergency Department at Fribourg Cantonal Hospital in Switzerland Using an Electronic TRIage Application: a Monocentric, Prospective Observational Study
Brief Title: FOllow-up of LOW-acuity Patients After REdirection From a Swiss Emergency Department Using an Electronic TRIage Application
Acronym: FO-LOW-RETRI
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Fribourgeois (Other)
Collaborators: University of Fribourg (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01655; HFR_24-09 (Other Grant/Funding Number: HFR-Fribourg)
Record Dates: First submitted 2025-03-19; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Triage; Low Acuity Patients; Health Literacy Level; Non-urgent Emergencies
Keywords: Patient Satisfaction; emergency department triage; patient redirection; healthcare system efficiency; Referral and Consultation; electronic decision support tool; patient flow; Emergency overcrowding
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Comparator Group (Current Practice - SETS-Based Triage and Redirection): * Patients are triaged using the Swiss Emergency Triage Scale (SETS)
  * Only low-acuity patients (SETS 4) are considered for redirection
  * Patients who agree to redirection are referred to external medical facilities (e.g., primary care clinics)
- Investigated Group (New Practice - Logibec-Assisted Triage and Redirection): * Patients tiraged as SETS 4 and SETS 3 are further evaluated by Logibec Réorientation software which applies applies specific inclusion/exclusion criteria to determine eligibility for redirection
  * Eligible patients are offered redirection, with appointments scheduled through the Reorientation software by the triage nurse
  Interventions: Other: intervention is the use of aTriage-Based Patient Redirection Using an Electronic Decision Support Toolin the emergency department (ED)

INTERVENTIONS:
Other: intervention is the use of aTriage-Based Patient Redirection Using an Electronic Decision Support Toolin the emergency department (ED) — Name: Logibec Réorientation software-assisted triage and redirection
  Type: Decision support system for emergency triage
  Implementation:
  * Applied during patient triage in the emergency department
  * Assists in identifying low-acuity (SETS 4) and semi-urgent (SETS 3) patients eligible for redirection
  * Uses standardized inclusion/exclusion criteria to guide redirection decisions
  Comparator: Standard nurse-led triage and redirection based only on the Swiss Emergency Triage Scale (SETS)
  Key Distinction:
  * The investigated group receives Logibec-assisted triage and redirection.
  * The comparator group follows traditional nurse-led triage without electronic support, limiting redirection to SETS 4 patients only.
  Groups: Investigated Group (New Practice - Logibec-Assisted Triage and Redirection)

SUMMARY:
Emergency department (ED) overcrowding is a growing issue, affecting patient safety, healthcare quality, and hospital efficiency. One strategy to manage low-acuity patients is triage-based redirection, where patients with non-urgent conditions are offered the option to receive care at external medical facilities instead of the ED.

This monocentric, prospective observational study will be conducted at Fribourg Cantonal Hospital, Switzerland, and evaluates the impact of a new electronic triage and redirection system (Logibec Réorientation). The study compares two triage processes:

Current practice - Redirection based on the Swiss Emergency Triage Scale (SETS), limited to low-acuity patients (SETS 4).

New practice - Redirection using the Logibec software, allowing redirection of both low-acuity (SETS 4) and semi-urgent (SETS 3) patients based on predefined criteria.

The primary objective is to assess whether the new triage-based redirection reduces the number of ED consultations per patient within 48 hours of their initial visit.

Secondary outcomes include:

Number of consultations in the ED or other medical facilities within 7 days Rate of hospital admissions within 7 days Patient satisfaction with redirection Evolution of health literacy over 6 months Number of ED visits over 6 months Participants are adult patients (≥18 years old) classified as SETS 3-4 and identified as eligible for redirection by the Logibec software. Data will be collected through phone interviews and questionnaires over a 6-month follow-up period.

This study aims to improve triage efficiency, patient flow management, and healthcare accessibility, while ensuring patient safety in the redirection process.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Triage level SETS 3 or SETS 4 (classified as semi-urgent or low-acuity)
* Identified as eligible for redirection by the Logibec electronic triage system
* Able to speak and read French or German (for informed consent and follow-up)
* Provides informed consent: Oral consent at Day 2 and Signed informed consent sent by post after inclusion

Exclusion Criteria:

* Inability to provide informed consent (e.g., cognitive impairment, language barrier without translation support)
* Inability to comply with study procedures, such as: Severe hearing impairment without hearing aids; Acute psychiatric conditions preventing participation; Not available for follow-up phone calls within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients (≥18 years old) seeking care at the Emergency Department (ED) of Fribourg Cantonal Hospital, Switzerland.
  This population consists of patients who:
  * present diverse medical complaints typically classified as with low-acuity (SETS 4) or semi-urgent (SETS 3) conditions as determined by the Swiss Emergency Triage Scale (SETS).
  * Are evaluated for potential redirection by ED triage nurse using the Logibec electronic triage system and may benefit from this triage-based redirection rather than hospital-based emergency care
  * Require non-urgent medical care that can be managed outside the hospital setting
  * French- or German-speaking individuals (for informed consent and follow-up participation)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Emergency Department Consultations per Patient Within 48 Hours After Initial Visit | From initial emergency department visit to 48 hours post-visit
  This measure refers to the total number of emergency department (ED) visits per patient within 48 hours following their initial presentation to the ED.
  The first consultation at the ED is counted as the initial visit.
  1. Any subsequent unplanned return visits to the ED within 48 hours of the initial visit are included in the count.
  2. Data collection is conducted through electronic health records (EHR) review and patient follow-up phone calls.
  This outcome aims to assess whether electronic triage-assisted redirection is effective, by providing service through alternative health care providers ,without patients needing further ED care

SECONDARY OUTCOMES:
the number of consultations per patient in the ED or other medical services within 7 days after the first ED visit | From initial emergency department visit to 7 days post-visit
the proportion of patients who need hospitalization related to initial complaint within 7 days | From initial emergency department visit to 7 days post-visit
the proportion of patients satisfied with the redirection process | At day 2 and day 7 post-visit
  Patient satisfaction as assessed by satisfaction questionnaire
the mean number of ED consultations after 1 month, 3 months and 6 months per patient | From initial emergency department visit to 6 month post-visit
the evaluation of the health literacy and its evolution within 6 months of visit | At day 7 post-visit and 6 months post-visit
  Health literacy as evaluated by EU-HLS-Q16 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ribordy, Prof., Study Director — HFR-Fribourg Emergency Department, University of Fribourg
Locations (1):
- HFR-Fribourg, Fribourg, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Due to patient confidentiality regulations, all data will be securely stored in a protected research database (REDCap), with access restricted to authorized study investigators. Only de-identified, aggregated results will be published in peer-reviewed journals and presented at scientific conferences. Identifiable patient information will not be shared outside the study team. Researchers may request summary-level data through formal collaboration agreements. This ensures compliance with data protection regulations while promoting scientific transparency.